CLINICAL TRIAL: NCT00083044
Title: Surrogate Endpoints in Prevention Studies and Ductal Lavage
Brief Title: Ductal Lavage in Assessing Women With Early Breast Cancer or at High Risk of Developing Breast Cancer and Who Are Eligible For Tamoxifen Therapy
Status: Withdrawn | Type: Observational
Why Stopped: Funding ended and will not be renewed
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: GRANT P50CA89018; NU-0649-003
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast cancer in situ; stage I breast cancer; lobular breast carcinoma in situ; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of or treat early cancer. Diagnostic procedures, such as ductal lavage, may improve the ability to assess the effectiveness of chemopreventive drugs, such as tamoxifen, on breast cells and may help doctors plan more effective treatment.

PURPOSE: This phase II trial is studying how well ductal lavage works in assessing changes in breast cells in women with early breast cancer or in those at high risk of developing breast cancer who are eligible for tamoxifen therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate cell morphology and protein expression of breast epithelial cells in ductal lavage samples as a marker of tamoxifen effect from women with breast cancer or from women at high risk for developing breast cancer.
* Evaluate methylation status of genes previously identified to be related to neoplastic progression of cells in ductal lavage samples from these participants.
* Evaluate the protein profile of nipple aspiration fluid from these participants before and after treatment with tamoxifen.

OUTLINE: This is a multicenter study.

Participants who are eligible for tamoxifen chemoprevention therapy undergo ductal lavage. Participants are informed of cytological findings and choose to receive oral tamoxifen once daily for 5 years vs observation only. All participants undergo repeat ductal lavage at 6 months. Participants with atypical cytology undergo a third ductal lavage at 12 months.

Mammographic density is measured at study entry and at 12 months.

Ductal cells are analyzed for methylation status of candidate genes.

Participants are followed as clinically indicated.

PROJECTED ACCRUAL: A total of 200 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of small invasive breast cancer
  * Diagnosis of ductal or lobular carcinoma in situ of the breast
  * At high risk for breast cancer (5-year Gail model risk of > 1.6%)
* Eligible for tamoxifen therapy
* No plans for adjuvant chemotherapy
* Prior unilateral early breast cancer allowed* NOTE: *Only the unaffected breast will be examined during this study
* Hormone-receptor status:

  * Estrogen receptor-positive (in patients with small invasive breast cancer)

PATIENT CHARACTERISTICS:

Age

* 18 to 64

Sex

* Female

Menopausal Status

* Premenopausal or postmenopausal

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No prior venous thromboembolism

Other

* At least 12 months post-partum
* Not pregnant
* Not nursing within the past 12 months
* No known allergy to lidocaine, prilocaine, or bupivacaine
* No uterine hyperplasia or polyps
* No other contraindication to tamoxifen

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 6 months since prior chemotherapy

Endocrine therapy

* Concurrent hormone-replacement therapy allowed
* Prior tamoxifen or raloxifene allowed provided treatment duration was no more than 6 months
* At least 1 year since prior raloxifene

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with early breast cancer or at high risk of developing breast cancer and who are eligible for tamoxifen therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Cell morphology and protein expression of breast epithelial cells in duct lavage samples as a marker of tamoxifen effect | Before and after tamoxifen treatment
Methylation status of genes previously identified to be related to neoplastic progression of cells in ductal lavage samples | At time of each ductal lavage.
Protein profile of nipple aspiration fluid before and after tamoxifen treatment | Before and after tamoxifen treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Seema A. Khan, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois

REFERENCES:
- [Background] Bhandare DJ, Khan SA, Motchoulskaia NA, Melnikov AA, Levenson Chernokhvostov VV. Isolation of highly purified DNA from low-abundance archived and stained cytological specimens. Clin Chim Acta. 2006 May;367(1-2):211-3. doi: 10.1016/j.cca.2005.12.022. Epub 2006 Feb 2. No abstract available. PMID 16458282
- [Background] Gorla SR, Steel J, Cohn R, et al.: Impact of surgical resection of primary breast tumor in stage IV breast cancer on local control and survival. [Abstract] J Clin Oncol 23 (Suppl 16): A-629, 35s, 2005.
- [Background] Li J, Zhao J, Yu X, Lange J, Kuerer H, Krishnamurthy S, Schilling E, Khan SA, Sukumar S, Chan DW. Identification of biomarkers for breast cancer in nipple aspiration and ductal lavage fluid. Clin Cancer Res. 2005 Dec 1;11(23):8312-20. doi: 10.1158/1078-0432.CCR-05-1538. PMID 16322290
- [Background] Golewale NH, Bryk M, Nayar R, et al.: Technical modifications of ductal lavage to improve cell yield. [Abstract] Breast Cancer Research and Treatment 82 (Suppl 1): A-1024, 2003.
- [Result] Patil DB, Lankes HA, Nayar R, Masood S, Bryk M, Hou N, Rademaker A, Khan SA. Reproducibility of ductal lavage cytology and cellularity over a six month interval in high risk women. Breast Cancer Res Treat. 2008 Nov;112(2):327-33. doi: 10.1007/s10549-007-9861-8. Epub 2007 Dec 21. PMID 18097749
- [Result] Fackler MJ, Malone K, Schilling E, et al.: Methylated genes in ductal lavage fluid from women with known breast cancer undergoing mastectomy. [Abstract] Breast Cancer Res Treat 94 (Suppl 1): A-2007, S85, 2005.
- [Result] Bhandare D, Bryk M, Nayar R, et al.: Effect of Tamoxifen (TAM) on estrogen-related biomarkers in ductal lavage (DL) samples a study on follow-up lavages. [Abstract] Breast Cancer Research and Treatment 88 (Suppl 1): A-4031, 2004.
- [Result] Bhandare D, Golewale N, Geiger A, et al.: Estrogen related biomarkers and cellular atypia in ductal lavage (DL) samples from women at high risk for breast cancer. [Abstract] Breast Cancer Res Treat 82 (Suppl 1): A-1032, S178, 2003.
- [Result] Didwania A, Golewale NH, Khan SA, et al.: Influence of ductal lavage (DL) findings on tamoxifen decision for high risk women. [Abstract] Breast Cancer Res Treat 82 (Suppl 1): A-1037, S179, 2003.